CLINICAL TRIAL: NCT02769481
Title: A Phase 3, Randomized, Double-blind, Active-controlled Study to Evaluate the Effects of Bexagliflozin Versus Glimepiride in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control by Metformin
Brief Title: Safety and Efficacy of Bexagliflozin Compared to Glimepiride as Add-on Therapy to Metformin in Type 2 Diabetes Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-1442-C-480
Record Dates: First submitted 2016-05-03; First posted 2016-05-11 (Estimated); Results first posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — bexagliflozin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bexagliflozin (Active Comparator): Subjects will receive a bexagliflozin tablet, 20 mg, once daily for the duration of the study. Subjects will continue taking metformin and receive placebo for glimepiride daily for the duration of the study.
  Interventions: Drug: Bexagliflozin; Drug: Placebo for Glimepiride
- Glimepiride (Active Comparator): Subjects will receive a glimepiride capsule, 2, 4 or 6 mg, once daily for the duration of the study. Subjects will continue taking metformin and receive placebo for bexagliflozin for the duration of the study.
  Interventions: Drug: Placebo for Bexagliflozin; Drug: Glimepiride

INTERVENTIONS:
Drug: Bexagliflozin — 20 mg, tablet
  Other Names: EGT0001442
  Arms: Bexagliflozin
Drug: Placebo for Bexagliflozin — inactive tablet to match active comparator bexagliflozin
  Arms: Glimepiride
Drug: Glimepiride — 2, 4 or 6 mg, capsule
  Arms: Glimepiride
Drug: Placebo for Glimepiride — inactive capsules to match active comparator glimepiride
  Arms: Bexagliflozin

SUMMARY:
The purpose of this study is to investigate the effect of bexagliflozin compared to glimepiride as an add-on therapy to metformin in lowering hemoglobin A1c (HbA1c) levels in subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Approximately 420 subjects with inadequately controlled T2DM on metformin will be recruited from North America and Europe. Subjects will be randomly assigned to receive bexagliflozin tablets, 20 mg, or glimepiride capsules, 2, 4 or 6 mg, in a ratio of 1:1 once daily for 96 weeks. Subjects will continue to take metformin for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM
* Currently taking metformin or taking metformin and one additional oral medication for diabetes
* Body Mass Index (BMI) ≤ 45 kg/m2
* Stable dose of blood pressure or cholesterol medications (if applicable) for at least 30 days

Exclusion Criteria:

* Hypersensitivity or other contraindication to the safe use of sulfonylurea or glimepiride
* Diagnosis of type 1 diabetes mellitus or maturity-onset/diabetes of the young
* Current use of injected therapy for treatment of diabetes (insulin or GLP-1 receptor agonist therapy) or thiazolidinedione class drugs
* History of genitourinary tract infections
* Evidence of abnormal liver function
* Myocardial infarction, stroke or hospitalization for heart failure within 3 months of screening
* Prior kidney transplant or evidence of kidney problems
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Paul Lock, MD, Study Director — Theracos Sub, LLC
Locations (45):
- United States (11):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntington Park, California
  - Research Site, Los Angeles, California
  - Research Site, San Carlos, California
  - Research Site, Hialeah, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Calabash, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Magnolia, Texas
- Germany (8):
  - Research Site, Aschaffenburg
  - Research Site, Essen
  - Research Site 2, Essen
  - Research Site 2, Hamburg
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Magdeburg
  - Research Site, Wangen
- Poland (16):
  - Research Site, Bochnia
  - Research Site, Bydgoszcz
  - Research Site, Krakow
  - Research Site 2, Krakow
  - Research Site, Lodz
  - Research Site 2, Lublin
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Puławy
  - Research Site, Staszów
  - Research Site, Swarzędz
  - Research Site, Świdnik
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Zamość
- Spain (10):
  - Research Site, Alicante
  - Research Site 2, Barcelona
  - Research Site, Barcelona
  - Research Site 2, Madrid
  - Research Site 3, Madrid
  - Research Site, Madrid
  - Research Site 2, Málaga
  - Research Site, Málaga
  - Research Site 2, Oviedo
  - Research Site, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bexagliflozin: Subjects will receive a bexagliflozin tablet, 20 mg, once daily for the duration of the study. Subjects will continue taking metformin and receive placebo for glimepiride for the duration of the study.
  Bexagliflozin tablets: 20 mg
  Glimepiride capsules: Placebo, inactive capsule to match the active comparator
- Glimepiride: Subjects will receive a glimepiride capsule, 2, 4 or 6 mg, once daily for the duration of the study. Subjects will continue taking metformin and receive placebo for bexagliflozin for the duration of the study.
  Bexagliflozin: Placebo, inactive tablet to match the active comparator
  Glimepiride capsules: 2, 4 or 6 mg
Period: Overall Study
Arm/Group | Bexagliflozin | Glimepiride
Started | 213 | 213
Study Complete at Week 60 | 193 | 192
Completed | 180 | 177
Not Completed | 33 | 36
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 3 | 6
Not completed — Entry Criteria Not Met | 1 | 2
Not completed — Withdrawal by Subject | 14 | 16
Not completed — Lost to Follow-up | 9 | 9
Not completed — Physician Decision | 0 | 1
Not completed — Terminated by Sponsor | 1 | 0
Not completed — Death | 0 | 1
Not completed — Undefined | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bexagliflozin | Glimepiride | Total
Number analyzed (Participants) | 213 | 213 | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.06) | 59.7 (10.35) | 59.6 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 83 | 178
  Male | 118 | 130 | 248
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 47 | 93
  Not Hispanic or Latino | 167 | 166 | 333
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 4 | 9
  White | 198 | 204 | 402
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 65 | 63 | 128
  Poland | 74 | 79 | 153
  Germany | 28 | 29 | 57
  Spain | 46 | 42 | 88
Height [Mean (Standard Deviation); unit: cm] | 166.7 (11.13) | 167.1 (9.53) | 166.9 (10.35)
Body Weight at Baseline [Mean (Standard Deviation); unit: kg] | 87.95 (19.122) | 90.23 (17.616) | 89.09 (18.399)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.45 (4.861) | 32.22 (5.155) | 31.83 (5.019)
Systolic Blood Pressure at Baseline [Mean (Standard Deviation); unit: mm Hg] | 133.3 (14.88) | 134.2 (14.37) | 133.8 (14.62)
Systolic Blood Pressure Categories [Count of Participants; unit: Participants]
  < 140 mm Hg | 135 | 138 | 273
  > 140 mm Hg | 78 | 75 | 153

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 60
Description: The primary objective is to demonstrate that bexagliflozin is non-inferior to glimepiride by evaluating the treatment effect on HbA1c reduction at week 60 in subjects whose T2DM is inadequately controlled by metformin. The least square mean (LSM) change from baseline to Week 60 was analyzed using a mixed model repeated measures (MMRM) analysis of covariance model (ANCOVA).
Time Frame: Baseline and Week 60
Population: The intention-to-treat population was used for the analysis. Subjects with a value at baseline and at week 60 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglin
Arm/Group | Bexagliflozin | Glimepiride
Number analyzed (Participants) | 193 | 191
percentage of glycated hemoglin | -0.70 (0.058) | -0.66 (0.058)
Statistical Analysis 1: Comparison: Bexagliflozin vs Glimepiride; The null hypothesis for the primary endpoint was that the change in HbA1c from baseline to week 60 in the bexagliflozin arm would be greater than change in the glimepiride arm by greater than 0.35%; Test type: Non-Inferiority — A 95% CI was to be calculated to estimate the range of values in which the treatment difference was likely to lie. If the 95% CI fell below the specified non inferiority margin of 0.35%, the non inferiority of bexagliflozin treatment to glimepiride treatment would be demonstrated and the null hypothesis would be rejected; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.21 to 0.11] — A lower value represents a better treatment effect

2. Secondary Outcome: Change From Baseline in Body Weight at Week 60 for Subjects With Baseline BMI ≥ 25 kg/m2
Description: Least squares (LS) mean treatment difference between the bexagliflozin group and placebo group in the change of body weight in subjects with baseline BMI ≥ 25 kg/m2 at week 60 is analyzed using ANCOVA.
Time Frame: Baseline and 60 weeks
Population: Number of subjects with a value at baseline and at the specified visit
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Bexagliflozin | Glimepiride
Number analyzed (Participants) | 182 | 182
kg | -3.71 (0.285) | 0.59 (0.284)
Statistical Analysis 1: Comparison: Bexagliflozin vs Glimepiride; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; Region, background treatment, baseline HbA1c, baseline eGFR, treatment, visit, treatment-by-visit and baseline weight as a fixed effect covariate; Difference of LS Means = -4.31, 95% CI 2-sided [-5.10 to -3.52]

3. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 60 for Subjects With Baseline SBP ≥ 140 mmHg
Description: Least squares (LS) mean treatment difference between the bexagliflozin group and placebo group in the change of SBP in subjects with baseline SBP ≥ 140 mmHg at week 60 is analyzed using ANCOVA.
Time Frame: Baseline and 60 weeks
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bexagliflozin | Glimepiride
Number analyzed (Participants) | 74 | 68
mm Hg | -13.48 (1.404) | -6.95 (1.460)
Statistical Analysis 1: Comparison: Bexagliflozin vs Glimepiride; Test type: Superiority; p = 0.0008, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 2, analysis 1]; Difference of LS Means = -6.53, 95% CI 2-sided [-10.56 to -2.51]

4. Secondary Outcome: Difference in Proportion of Subjects With ≥ 1 Severe or Documented Symptomatic Hypoglycemia Events Over 96 Weeks
Description: The difference in proportion of subjects with ≥ 1 severe or documented symptomatic hypoglycemia events in the bexagliflozin group compared with glimepiride group over 96 weeks is analyzed using a logistic regression model. The full model included region, baseline HbA1c value, background treatment status (metformin or metformin + OHA), eGFR at baseline ≥ 90 or < 90 mL min 1 per 1.73 m2), treatment as a fixed effect covariate.
Time Frame: During the 96 week treatment period
Population: Subjects with post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Bexagliflozin | Glimepiride
Number analyzed (Participants) | 213 | 212
Proportion of participants | 0.02 [0.01 to 0.05] | 0.15 [0.10 to 0.22]
Statistical Analysis 1: Comparison: Bexagliflozin vs Glimepiride; Test type: Superiority; p < 0.0001, Regression, Logistic — P-value is based on one sided statistical tests using a 0.025 level of significance; Region, baseline HbA1c, background treatment, eGFR at baseline, treatment as a fixed effect covariate; Odds Ratio (OR) = 0.12, 95% CI 2-sided [0.05 to 0.28] — Odds ratio is calculated as the odds ratio of bexagliflozin over glimepiride

5. Secondary Outcome: Superiority of Bexagliflozin Over Glimepiride in HbA1c Reduction at Week 60.
Description: Superiority of bexagliflozin over glimepiride in HbA1c reduction from baseline to week 60 will be declared if the upper bound of 95% CI is less than 0.
Time Frame: Baseline to Week 60
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Bexagliflozin | Glimepiride
Number analyzed (Participants) | 193 | 191
percentage of glycated hemoglobin | -0.70 (0.058) | -0.66 (0.058)
Statistical Analysis 1: Comparison: Bexagliflozin vs Glimepiride; Test type: Superiority — Superiority of bexagliflozin over glimepiride in HbA1c reduction from baseline to week 60 will be declared if the upper bound of 95% confidence interval is less than 0; Difference of LS Means = -0.05, 95% CI 2-sided [-0.21 to 0.11]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Week -8 (V2, wash-out) to Week 98 (V18, follow-up).
Arm/Group | Bexagliflozin | Glimepiride
All-Cause Mortality (participants affected / at risk) | 0/213 | 1/213
Serious Adverse Events (participants affected / at risk) | 25/213 | 26/213
Other Adverse Events (participants affected / at risk) | 98/213 | 112/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bexagliflozin (N=213) | Glimepiride (N=213)
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Myocardial ischemia (Cardiac disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Palpitation (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Erysipelas (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischemic stroke (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Thalamic infarction (Nervous system disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Contusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle rupture (Musculoskeletal and connective tissue disorders) | 1 | 0
Tibia fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Ectropion (Eye disorders) | 1 | 0
Entropion (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Bladder disorder (Renal and urinary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Genital hemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bexagliflozin (N=213) | Glimepiride (N=213)
Hypoglycemia (Metabolism and nutrition disorders) | 36 | 71
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 17
Nasopharyngitis (Infections and infestations) | 29 | 29
Urinary Tract Infection (Infections and infestations) | 25 | 10
Bronchitis (Infections and infestations) | 14 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator has no publication right.

DOCUMENTS (2):
  • Study Protocol (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT02769481/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT02769481/SAP_001.pdf